CLINICAL TRIAL: NCT01422980
Title: Effect of Consumption of Dairy Product on Upper Gastric Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU345
Record Dates: First submitted 2011-04-21; First posted 2011-08-25 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Upper Gastric Discomfort
Keywords: dairy product; upper gastric discomfort; adult

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Test product (Active Comparator): Arm 1 - intervention 1 (test product)
  Interventions: Other: 1- Test dairy product containing specific ingredients
- 2 = Control product (Placebo Comparator): Arm 2 - intervention 2 (control product)
  Interventions: Other: 2- Control dairy product without specific ingredients

INTERVENTIONS:
Other: 1- Test dairy product containing specific ingredients
  Arms: 1 = Test product
Other: 2- Control dairy product without specific ingredients
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to determine whether the consumption of test dairy products is effective in reducing upper gastric discomfort after 2 weeks of product consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 21 - 60 years old
* Experiencing upper gastric discomfort

Exclusion Criteria:

* Participants with alarm symptoms (dysphagia, bleeding, involuntary weight loss clinically significant >10% of it habitual weight during the last 6 months).
* Participants with diagnosed severe organic esophageal medical history (endoscopic eosophagitis A, B, C or D of Los Angeles classification, peptic stenosis, Barrett oesophagus, huge hiatus hernia or para-esophageal) gastric or duodenal ulcer or high digestive haemorrhage clinical history.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in gastro-oesophageal symptoms as assessed by RDQ questionnaire | Two timepoints are considered in the assessment of the change outcome measures: from Baseline (before product consumption) to Endpoint (i.e. final evaluation visit after 2 weeks of product consumption)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano, Buenos Aires, Argentina